CLINICAL TRIAL: NCT04717635
Title: An Open-label, Single-arm, Active-treatment Study to Evaluate Efficacy and Safety of Canakinumab (ACZ885) Administered for at Least 48 Weeks in Japanese Patients With Adult Onset Still's Disease (AOSD)
Brief Title: Study of Efficacy and Safety of Canakinumab in Japanese Patients With AOSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885G1302; 2021-003706-50 (EudraCT Number)
Record Dates: First submitted 2020-12-18; First posted 2021-01-22 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Adult Onset Still's Disease
Keywords: Canakinumab; AOSD; IL-1β; Japanese participants
MeSH Terms: conditions — Still's Disease, Adult-Onset | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canakinumab (Experimental): All participants receive canakinumab (ACZ885) as open-label study medication. Participants are administered canakinumab 4 mg/kg every 4 weeks. The maximal total single dose of canakinumab allowed is 300 mg.
  Interventions: Biological: Canakinumab

INTERVENTIONS:
Biological: Canakinumab — Provide as 150 mg/1 mL solution for subcutaneous injection and administer 4mg/kg every 4 weeks.
  Other Names: ACZ885

SUMMARY:
This is a phase III study designed to provide efficacy and safety data for canakinumab administered for at least 48 weeks as subcutaneous (s.c.) injection every 4 weeks (q4wk) in Japanese patients with Adult Onset Still's Disease (AOSD). Interim analysis (IA) data at Week 28 and 48 from this study supports a registration submission of canakinumab in the indication of Adult still's disease (ASD) in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study. Parent's or legal guardian's written informed consent and child's assent, if appropriate, are required before any assessment is performed for participants < 20 years of age
* Japanese male and female participants aged ≥ 16 years
* Confirmed diagnosis of AOSD as per Yamaguchi criteria (Yamaguchi M, 1992) with an onset of disease ≥ 16 years of age. Yamaguchi criteria requires at least five criteria, including two major criteria and no exclusion criteria
* Active disease at the time of baseline defined as follows
* Fever (body temperature > 38°C) due to AOSD for at least 1 day within 1 week before baseline
* At least 2 active joints (tender or swollen)
* CRP ≥ 10 mg/L

Exclusion Criteria:

* Pregnant or nursing (lactating) female participants, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/ mL) at screening visit.
* History of significant hypersensitivity to study drug or to biologics.
* History/evidence of active macrophage activation syndrome or disseminated intravascular coagulation prior to 6 months of enrollment.
* With underlying metabolic, renal, hepatic, infectious or gastrointestinal conditions which in the opinion of the investigator compromises the articipant and/ or places the participant at unacceptable risk for participation in an immunomodulatory therapy.
* With active or recurrent bacterial, fungal or viral infection at the time of enrollment, including participants with evidence of Human Immunodeficiency Virus (HIV) infection, Hepatitis B and Hepatitis C infection.
* Participants with absolute neutrophil count < 1500/mm3 at screening.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve adapted American College of Rheumatology (ACR) 30 response at Week 8 | Week 8
  Adapted ACR30 response is defined as 30% reduction between baseline and post-baseline values in at least 3 of the 5 response variables 1 to 5 and no intermittent fever in the preceding week (variable 6), with no more than one of variables 1-5 worsening by more than 30%:
  1. Physicians global assessment of disease activity
  2. Participant's assessment of disease activity (PtGA)
  3. Functional ability assessed using Health Assessment Questionnaire (HAQ)
  4. Number of active joints (68 joints evaluated for pain/tenderness and 66 for swelling)
  5. Laboratory measure of inflammation: CRP (mg/L)
  6. Absence of intermittent fever in the preceding week

SECONDARY OUTCOMES:
Proportion of participants who are able to taper corticosteroids based on success criteria at Week 28. | Week 28
  To evaluate ability of canakinumab to taper corticosteroids based on success criteria starting from Week 8 to Week 28
Proportion of participants who achieved adapted ACR 30/50/70/90/100 response criteria at Day 15 and all subsequent visits. | Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, End of Study(EOS)(up to Week 152)
  The adapted ACR 50, 70, 90 and 100 criteria will be used as additional efficacy assessments, i.e., an improvement ≥ 50%, ≥ 70%, ≥ 90%, or = 100% in at least 3 of 5 response variables and no intermittent fever in the preceding week (variable 6) with no more than one variable of 1-5 worsening by more than 30%.
Change from baseline in Systemic Feature Score (total score and each components) at Day 15 and all subsequent visits. | Baseline, Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, EOS(up to Week 152)
  Systemic feature score consists of 5 clinical and 5 laboratory assessments. Clinical features include fever, rash, lymphadenopathy, hepatosplenomegaly and serositis. Laboratory features include erythrocyte sedimentation rate, C reactive protein, leucocyte count, hemoglobin level and platelet count. Each clinical and laboratory feature will be assigned a score of 1 (present) or 0 (absent):
Absolute change from baseline in the component of adapted ACR at Day 15 and all subsequent visits: Physician's global assessment of disease activity | Baseline, Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, EOS(up to Week 152)
  The physician will rate the participant's current condition on a 0-100 mm Visual Analog Scale (VAS), ranging from no disease activity (0 mm) to very severe disease activity (100 mm).
Absolute change from baseline in the component of adapted ACR at Day 15 and all subsequent visits: Patient's global assessment of disease activity | Baseline, Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, EOS(up to Week 152)
  The participant's assessment of disease activity will be assessed on the VAS. The VAS scale ranges from 0-100 mm, from no pain/very well (0 mm) to very severe pain/very poor (100 mm).
Absolute change from baseline in the component of adapted ACR at Day 15 and all subsequent visits: Health Assessment Questionnaire | Baseline, Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, EOS(up to Week 152)
  The health assessment questionnaire, HAQ©, will be used to assess physical ability and functional status of participants as well as quality of life. The disability dimension consists of 20 multiple choice items concerning difficulty in performing eight common activities of daily living; dressing, arising, eating, walking, hygiene, reach, grip and usual activities. Participants choose from four response categories, ranging from 'without any difficulty' to 'unable to do'.
Absolute change from baseline in the component of adapted ACR at Day 15 and all subsequent visits: Tender and swollen joint counts | Baseline, Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, EOS(up to Week 152)
  Active joints are defined as joints with swelling or pain/tenderness. 68 joints will be assessed for tenderness and 66 joints for swelling.
Absolute change from baseline in the component of adapted ACR at all visits: C-Reactive Protein(CRP) | Baseline, Days 3, 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, 112, 116, 120, 124, 128, 132, 136, 140, 144, 148, EOS(up to Week 152)
  CRP values were standardized to a normal range of 0 to 10 mg/L.
Absolute change from baseline in the component of adapted ACR at all visits: Fever assessment | Baseline, Days 3, 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, 112, 116, 120, 124, 128, 132, 136, 140, 144, 148, EOS(up to Week 152)
  The absence or presence of intermittent fever due to AOSD (oral, rectal, or axillary body temperature > 38°C only for several hours during the day) will be assessed.
Change from baseline of corticosteroid dose at all visits after Week 8. | Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, 112, 116, 120, 124, 128, 132, 136, 140, 144, 148, EOS(up to Week 152)
  To evaluate ability of canakinumab to taper corticosteroids dose over time after Week 8
Presence of rash (typical/atypical) at all visits during study. | Baseline, Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, 112, 116, 120, 124, 128, 132, 136, 140, 144, 148, EOS(up to Week 152)
  The absence or presence of skin rash will be assessed based on physical exam findings including whether it is typical or atypical.
Change from baseline in DAS28-CRP at Day 15 and all subsequent visits. | Baseline, Day 15, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, EOS(up to Week 152)
  DAS28-CRP is a composite index, validated for RA patients and takes into account the following items: Tender joint count (number of tender joints; 0-28); swollen joint count (number of swollen joints; 0-28); C-reactive protein (mg/l) and Global Health (Patient's Global Assessment of Disease Activity; from 0=best to 100=worst). Thus, given the reliability, validity, and ability of DAS28 to discriminate the severity of joint involvement, this index has been used in other rheumatic diseases characterized by RA-like poly-articular involvement. Of note, a DAS28 score > 5.1 implies active disease, ≤3.2 low disease activity, and <2.6 remission. Moderate/high disease activity is defined as a DAS28 higher than 3.2.
Canakinumab concentrations over time | Baseline, Days 3, 15, Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  To evaluate the pharmacokinetics (PK) of canakinumab
Total IL-1β (sum of IL-1β free and bound to canakinumab) level s over time | Baseline, Days 3, 15, Weeks 4, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  To evaluate the pharmacodynamic (PD) of canakinumab
Anti-canakinumab antibody identification and titer | Baseline, Weeks 24, 48, 72, 96, 120
  To assess the immunogenicity of canakinumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Japan (9):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chiba

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com